CLINICAL TRIAL: NCT01938131
Title: Effectiveness of Treatment With rMV (Repeated Muscle Vibration) in Patients Affected by Knee Osteoarthritis: a Prospective Randomized Clinical Trial
Brief Title: Study of Effectiveness of rMV (Repeated Muscle Vibration) in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Carlo Bertolini, Principal Investigator, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1346/2012
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Knee Osteoarthritis
Keywords: knee, osteoarthritis, muscle vibration
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Patients in this group will be subjected to a treatment with muscle released in which the probe of CroSystem instrument will be approached to the quadriceps, without making contact. The instrument in these conditions emits a buzz but not provokes muscle vibration
- repeated Muscle Vibration (Experimental): The patients will be subjected to 3 daily applications of rMV of 10 minutes each, for 3 consecutive days. Between two successive applications will be observed a break of at least 15 seconds. The probe of the specific instrument (Cro ® System) will be placed near the supero-medial margin of the patella, on both quadriceps
  Interventions: Device: repeated Muscle Vibration (rMV) (Cro ® System)

INTERVENTIONS:
Device: repeated Muscle Vibration (rMV) (Cro ® System) — The patients will be subjected to 3 daily applications of rMV of 10 minutes each, for 3 consecutive days. Between two successive applications will be observed a break of at least 15 seconds. The probe of the specific instrument (Cro ® System) will be placed near the supero-medial margin of the patella, on both quadriceps
  Arms: repeated Muscle Vibration

SUMMARY:
The rehabilitation protocols in knee osteoarthritis are often difficult to be applied in elderly patients because they are long lasting and need the constant participation of patients. To rapidly improve the motor performances of patients it is possible to use the mechanical vibration applied to individual muscles using a protocol called "repeated muscle vibration" (rMV). The purpose of this single-blind randomized placebo-controlled study is to evaluate the effectiveness of the repeated muscle vibration (rMV) in terms of increasing the ability of the patients affected by knee osteoarthritis, compared to an ineffective treatment, considered as a placebo. Each subject, randomly assigned to either the group 1 (study group) or placebo-treatment (group 2)is administered 3 daily applications of rMV of 10 minutes each, for 3 consecutive days. Between two successive applications it's observed a break of at least 15 seconds. The probe of the specific instrument (Cro ® System) is placed near the supero-medial margin of the patella, on both quadriceps. Patients in group 2 (control group) are subjected to a treatment with muscle released in which the probe of the same instrument is approached to the quadriceps, without making contact. The instrument in these conditions emits a buzz but not provokes muscle vibration. The primary outcome of the study is to determine the changing in patients' ability (as measured by WOMAC scale = Western Ontario and McMaster Universities Osteoarthritis Index) . The secondary outcomes of the study are the assessment of changing of patients' balance and risk of falling (as measured by the Tinetti scale) and assessment of changing of patients' quality of life (as measured by EQ-VAS= EuroQuality of Life-VAS scale).Outcome measures are administered at baseline (T0), at the end of the treatment protocol (T1), at 1 month (T2), 3 months (T3) after the end of treatment and 6 months (T4) after the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Knee Osteoarthritis

Exclusion Criteria:

* Neurologic disease involving the lower limbs or causing balance problems
* Systemic inflammatory diseases
* Diabetic Neuropathy
* Severe heart disease.
* Acute infections or bone Tuberculosis
* Prosthetic lower limbs
* History of surgery on the affected knee in the last year
* History of cancer
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
changing in patients' ability (as measured by WOMAC scale) | baseline (T0), at the end of the treatment protocol (T1), at 1 month (T2), 3 months (T3) after the end of treatment, 6 months (T4) after the end of the treatment
  administration of WOMAC scale for patient's ability evaluation

SECONDARY OUTCOMES:
assessment of changing of patients' balance and risk of falling (as measured by the Tinetti scale) | baseline (T0), at the end of the treatment protocol (T1), at 1 month (T2), 3 months (T3) after the end of treatment, 6 months (T4) after the end of the treatment
  administration of Tinetti scale for patient's balance and risk of falling evaluation
assessment of changing of patients' quality of life (as measured by EQ-VAS) | baseline (T0), at the end of the treatment protocol (T1), at 1 month (T2), 3 months (T3) after the end of treatment, 6 months (T4) after the end of the treatment
  administration of EQ-VAS scale for patient's pain evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital "A. Gemelli", Catholic University of the Sacred Heart, Rome, Italy, Italy